CLINICAL TRIAL: NCT01706419
Title: Fortified Rice for School Children in Cambodia: Effects on Micronutrient Status, Growth, Cognition and Health.
Brief Title: Fortified Rice for School Children in Cambodia
Acronym: FORISCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Department of Fisheries Post-harvest Technologies and Quality Control (Other); World Food Program Cambodia (Unknown); PATH (Other)
Responsible Party: Principal Investigator, Frank Wieringa, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FORISCA
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Micronutrient Status
Keywords: vitamin A; iron; zinc; school children; fortified rice; morbidity; growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- no school meal (No Intervention): control group receiving no school meal
- normal school meal (Placebo Comparator): school meal without fortified rice, placebo group
- cold extruded fortified rice (Experimental): school meal with fortified rice using cold extrusion kernels
  Interventions: Dietary Supplement: Fortified rice cold extruded kernel
- warm extrusion (Experimental): school meal with fortified rice using warm extrusion kernels
  Interventions: Dietary Supplement: fortified rice warm extruded kernel
- hot extruded (Experimental): school meal with fortified rice using hot extrusion kernels
  Interventions: Dietary Supplement: fortiified rice hot extruded kernel

INTERVENTIONS:
Dietary Supplement: Fortified rice cold extruded kernel
  Arms: cold extruded fortified rice
Dietary Supplement: fortified rice warm extruded kernel
  Arms: warm extrusion
Dietary Supplement: fortiified rice hot extruded kernel
  Arms: hot extruded

SUMMARY:
Rice fortification has been shown to be safe and effective in improving micronutrient status in many studies around the world. However, most studies have been done in Latin America, Africa and India. There are no studies available from Cambodia. Moreover, there is no data available on whether fortified rice can reduce the prevalence of anemia in school children in Cambodia, nor whether there will be additional benefits, such as better learning capability of school children or fewer days missed due to better health. To inform WFP, Cambodian policy and the public on the potential benefits of fortified rice on health and development for Cambodian school children, an intervention study will be conducted in Kampung Speu province during the 2012 - 2013 school year. The study will be conducted by IRD, PATH and WFP. Sixteen schools will be selected to receive either the normal rice provided by the WFP school meal program, or fortified rice instead of normal rice. Three (3) different types of fortified rice will be tested, to identify the best type of fortified rice. In addition, 4 schools with no school meal program will be selected to serve as control. School attendance and morbidity will be followed in all children in the participating schools over the whole school year. Biochemical indicators of micronutrient status will be determined in a subgroup of children (25% of the children), which requires collection of blood, urine and stool samples.

DETAILED DESCRIPTION:
Micronutrient deficiencies are a major health problem in many developing countries, including Cambodia. Micronutrient deficiency results in poor health, with a much higher risk for mortality in vulnerable groups such as pregnant women and young infants, and delayed physical and cognitive development, resulting in retarded growth and stunting. It thereby prevents children from reaching their full potential as micronutrients play an important role in children's cognitive and motor development.

The UN World Food Program (WFP) provides a daily school meal to ~500,000 school children in Cambodia. The main objective of the school meal program is to increase school attendance. Although the school meal provides salt fortified with iodine, and vegetable oil fortified with vitamin A, the school meal provides an excellent opportunity to improve micronutrient status of school children by providing them with rice fortified with vitamins and minerals such as zinc, vitamin A, iron, folic acid and vitamin B12. This is likely to reduce the prevalence of anemia in school children and improve health and school performance. Anemia is a major problem in school children in Cambodia. A recent study by WFP showed that more than half of the school children were anemic.

Rice fortification has been shown to be safe and effective in improving micronutrient status in many studies. However, most studies have been done in Latin America, Africa and India. There are no studies available from Cambodia, except for an acceptability study of fortified rice conducted by WFP and the Institute of Research for Development (IRD) in 2010 in Kampung Speu. This acceptability study showed that fortified rice has an excellent acceptability among school children, parents and teachers. However, there is no data available on whether fortified rice can reduce the prevalence of anemia in school children in Cambodia, nor whether there will be additional benefits, such as better learning capability of school children or fewer days missed due to better health.

To inform WFP, Cambodian policy and the public on the potential benefits of fortified rice on health and development for Cambodian school children, an intervention study will be conducted in Kampung Speu province during the 2012 - 2013 school year. The study will be conducted by IRD, PATH and WFP. Sixteen (16) schools will be selected to receive either the normal rice provided by the WFP school meal program, or fortified rice instead of normal rice. Three (3) different types of fortified rice will be tested, to identify the best type of fortified rice. In addition, 4 schools with no school meal program will be selected to serve as control. School attendance and morbidity will be followed in all children in the participating schools over the whole school year. Biochemical indicators of micronutrient status will be determined in a subgroup of children (25% of the children), which requires collection of blood, urine and stool samples.

The study will be submitted to the Ethical Committee of the Ministry of Health for approval, and the Ethical Review Board of PATH, USA. Furthermore, approval will be obtained from the Ministries of Health, Education and Planning prior to the commencement of the study.

Potential benefits of the study includes the immediate treatment of school children found to have severe anemia (hemoglobin < 70 g/L) and improved health and cognitive development for all children receiving fortified rice. Potential disadvantages and risks of the study include side effects of blood taking in the subgroup of children and the disruption of classes for a few days during the data collection.

If the results of the study show improved health and cognition for school children receiving fortified rice, provision of fortified rice to all 500,000 Cambodian school children taking part in the WFP school meal program in Cambodia could become a priority.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by parent / caretaker
* age between 6 and 14 yrs
* visiting selected school
* taking part in school meal program

Exclusion Criteria:

* any chronic illness affecting growth (such as HIV)
* no informed consent
* severe anemia which will require direct treatment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9500 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Anthropometry | 6 months
  Weight, height and skinfold thickness
Micronutrient status | 6 months
  iron, zinc, iodine and vitamin A status using plasma and urine concentrations
Cognition | 6 months
  Raven's colored matrices test and WISC III tests
absentism | 6 months
  days out of class
morbidity | 6 months
  days and number of episodes ill

SECONDARY OUTCOMES:
Parasite infestation | 6 months
  number of parasite eggs in stools
gut inflammation | 6 months
  calprotectin concentrations in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Frank T Wieringa, MD PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (1):
- Department of Fisheries Post-harvest Technologies and Quality Control, Fisheries Administration, Phnom Penh, Cambodia

REFERENCES:
- [Derived] Seyoum Y, Greffeuille V, Kouadio DKD, Kuong K, Turpin W, M'Rabt R, Chochois V, Fortin S, Perignon M, Fiorentino M, Berger J, Burja K, Ponce MC, Chamnan C, Wieringa FT, Humblot C. Faecal microbiota of schoolchildren is associated with nutritional status and markers of inflammation: a double-blinded cluster-randomized controlled trial using multi-micronutrient fortified rice. Nat Commun. 2024 Jun 18;15(1):5204. doi: 10.1038/s41467-024-49093-4. PMID 38890302
- [Derived] de Gier B, Campos Ponce M, Perignon M, Fiorentino M, Khov K, Chamnan C, de Boer MR, Parker ME, Burja K, Dijkhuizen MA, Berger J, Polman K, Wieringa FT. Micronutrient-Fortified Rice Can Increase Hookworm Infection Risk: A Cluster Randomized Trial. PLoS One. 2016 Jan 6;11(1):e0145351. doi: 10.1371/journal.pone.0145351. eCollection 2016. PMID 26735845